CLINICAL TRIAL: NCT03458169
Title: Usability of a New Overground Body Weight Support Rehabilitation Robot LEAP: A Monocentric Consideration-of-concept Trial
Brief Title: LEAP a New Overground Body Weight Support Robot: Usability Trial
Acronym: LEAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Romande de Readaptation (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CliniqueRR-05
Record Dates: First submitted 2017-12-21; First posted 2018-03-08 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2018-03

CONDITIONS: Spinal Cord Injuries; Cerebral Palsy; Parkinson Disease; Multiple Sclerosis; Stroke; People With Impaired Lower Extremity Function
MeSH Terms: conditions — Spinal Cord Injuries; Cerebral Palsy; Parkinson Disease; Multiple Sclerosis; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LEAP usability (Experimental): * Therapist LEAP session feedback
  * Participant LEAP session feedback
  * LEAP risk control validation
  Interventions: Device: Therapist LEAP session feedback; Device: Participant LEAP session feedback; Device: LEAP risk control validation

INTERVENTIONS:
Device: Therapist LEAP session feedback — A standard therapy session is being performed with a participant with the LEAP body-weight support robot. Subsequently, the therapist is answering a questionnaire to assess the clinical applicability of the robot. An observer will assess with a questionnaire whether use errors occurred during the session.
Device: Participant LEAP session feedback — A standard therapy session is being performed with a participant inside the LEAP body-weight support robot. Subsequently, the participant is answering a questionnaire to assess the comfort of the robot.
Device: LEAP risk control validation — The therapist rates the risk control measurements of the LEAP robot with a questionnaire, during a session with a member of the investigational team.

SUMMARY:
People with central nervous system disorders such as spinal cord injury, stroke, cerebral palsy, Parkinson's disease, multiple sclerosis, etc… often have impaired lower extremity function that limits activities of daily life and independence. Different body-weight support systems have been developed to facilitate the rehabilitation process by compensating for the user's residual abilities. However, studies on weight-supported gait training on a treadmill have failed to show superiority over conventional rehabilitation programs for spinal cord injury and stroke. A recent study by the group around Grégoire Courtine showed that body-weight support systems that provide assistance only in the vertical direction disrupt the production of gait and balance, suggesting that current practices may even be detrimental for relearning to walk. For the past year, the Clinique Romande de Réadaptation (CRR) worked together with the G-Lab at EPFL and G-Therapeutics on a new robot platform specifically developed to provide adjustable trunk support along four independent degrees of freedom (LEAP). The investigators were able to draw on their long-term experience, which consists of different body weight support training systems for stroke and spinal cord injury. This knowledge, combined with the input of our therapists and physicians and the specific requirements for people with neurological/musculoskeletal disorders, has resulted in a design that can provide adjustable bodyweight support during over-ground locomotion, treadmill, stairs training, standing up and sitting down and for support during the training of activities of daily living.

The scope of this study is to examine how well the robot can be used for rehabilitation therapy in everyday clinical practice. This includes, among other things, technical aspects such as the handling of the hardware, the adaptability of the robot to the patient, and the safety during operation (such as the fall prevention). Various patient-specific aspects will also be evaluated e.g. comfort, positioning, or motivation of the patient. This study also aims to evaluate the software with the various support modes, operating options, and the user interface of the LEAP.

ELIGIBILITY:
Healthy participants fulfilling all of the following inclusion criteria are eligible for the study:

* The healthy volunteer or legal representative has been informed and has signed the informed consent form
* Age 18-80 or age 5-10 (women or men)
* Weight below 137 kg
* Height between 120 and 190 cm
* Agree to comply in good faith with all conditions of the study and to attend all required training

Patients fulfilling all of the following inclusion criteria are eligible for the study:

* The patient has been informed and has signed the informed consent form
* Age 18-80 (women or men)
* Weight below 137 kg
* Height between 120 and 190 cm
* Neurological/musculoskeletal diagnoses
* Impairment of the lower extremities
* Stable medical and physical condition as considered by the attending doctor or physician
* Agree to comply in good faith with all conditions of the study and to attend all required training
* Other (non-neurological) diagnoses, who require intense training of the lower extremities
* The rehabilitation physician or doctor provides a final agreement whether the participant can train with the LEAP

The presence of any one of the following exclusion criteria will lead to exclusion of the participant, for example:

* Strong adipositas, which makes it not possible to adjust the harness to the anthropometrics of the participant
* Bracing of the spinal column.
* Severe joint contractures disabling or restricting lower limb movements
* Instabilities of bones or joints, fractures or osteoporosis/osteopenia
* Allergy against material of harness
* Open skin lesions
* Luxations or subluxations of joints that should be positioned in LEAP
* Strong pain
* Strong spontaneous movements like ataxia, dyskinesia, myoclonus*
* Instable vital functions like pulmonal or cardiovascular conditions
* Uncooperative or aggressive behaviour
* Severe cognitive deficits
* Inability to signal pain or discomfort
* Apraxia*
* Severe spasticity (Ashworth 4)
* Severe epilepsy*
* Insufficient head stability
* Infections requiring isolation of the patient
* History of significant autonomic dysreflexia
* Systemic malignant disorders
* Cardiovascular disorders restricting physical training
* Peripheral nerve disorders
* Other anatomic or co-morbid conditions that, in the investigator's opinion, could limit the patient's ability to participate in the study or to comply with follow-up requirements, or impact the scientific soundness of the study results.
* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Participation in another study with investigational drug within the 30 days preceding and during the present study
* Previous enrolment into the current study Contraindications marked with an * are relative contraindications. Final approval needs to be obtained from the attending medical doctor.

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Usability of the robot - Fixation | 2 minutes
  From the user/therapist the information on the usability of the robot (CRF I) is being assessed. This questionnaire is only filled once by each user/therapist.
  Feedback on patient/subject fixation (Ordinal scale from 1:useful to 5:not useful)
Usability of the robot - Applicability | 2 minutes
  From the user/therapist the information on the usability of the robot (CRF I) is being assessed. This questionnaire is only filled once by each user/therapist.
  Feedback on clinical applicability (Ordinal scale from 1:useful to 5:not useful)
Usability of the robot - Robot support | 2 minutes
  From the user/therapist the information on the usability of the robot (CRF I) is being assessed. This questionnaire is only filled once by each user/therapist.
  Feedback on robot support (Ordinal scale from 1:useful to 5:not useful)
Usability of the robot - User interface | 2 minutes
  From the user/therapist the information on the usability of the robot (CRF I) is being assessed. This questionnaire is only filled once by each user/therapist.
  Feedback on user interface (Graphical user interface) (Ordinal scale from 1:useful to 5:not useful)
Usability of the robot - Interaction | 2 minutes
  From the user/therapist the information on the usability of the robot (CRF I) is being assessed. This questionnaire is only filled once by each user/therapist.
  Feedback on the LEAP interaction (Ordinal scale from 1:useful to 5:not useful)
Risk control validation - Observer | 1 hour
  From an independent observer (investigator, or a member of the development team) the occurrence of use errors is recorded (CRF III):
  Each primary operating function of the robot is rated (Ordinal scale from 0 to 1 for 'use error occurred' or 'no use error' This questionnaire has only to be filled out once for each user/therapist.
Risk control validation - User | 1 hour
  The risk control measures are validated by the user/therapist (CRF IV):
  The different risk controls are rated (Ordinal scale from 0 to 1 for 'Acceptable' or 'Not acceptable') This questionnaire has only to be filled out once by each user/therapist.
Participant feeling of safety/comfort - Fixation | 1 minute
  From the participant information on the comfort/safety is being assessed (CRF II):
  Feedback on the fixation of the patient (Open-ended question)
Participant feeling of safety/comfort - Robot training | 1 minute
  From the participant information on the comfort/safety is being assessed (CRF II):
  Feedback on the robot training (Ordinal scale from 0 to 5)
Participant feeling of safety/comfort - Robot support | 1 minute
  From the participant information on the comfort/safety is being assessed (CRF II):
  Feedback on the robot support (Ordinal scale from 0 to 5)

SECONDARY OUTCOMES:
Robot Measurement - Patient position | 1 hour
  The robot records the patient position in the room (in meters).
Robot Measurement - Walking speed | 1 hour
  The robot records the walking speed (in meters per second).
Robot Measurement - Occurred errors | 1 hour
  The robot records the errors occurred (error number).
Robot Measurement - Support forces | 1 hour
  The robot records the support forces (in Newton).
Robot Measurement - Fall detection | 1 hour
  The robot records the number of detected falls (Amount of detected falls).
Robot Measurement - Walked distance | 1 hour
  The robot records the distance the patient walked during the session (in meters).
EMG system | 1 hour
  Upon availability, an EMG system will be used to measure muscle activity during the session.
Patient characteristics - Testing date | 1 minutes
  The testing date (day/month/year) is being recorded.
Patient characteristics - Identification number | 1 minutes
  A unique participant identification number is being recorded.
Patient characteristics - Body height | 1 minutes
  The body height (in cm) is being recorded.
Patient characteristics - Body weight | 1 minutes
  The body weight (in kg) is being recorded.
Patient characteristics - Waist size | 1 minutes
  The waist size (in cm) is being recorded.
Patient characteristics - Tight circumference | 1 minutes
  The tight circumference (in cm) is being recorded.
Patient characteristics - Chest size | 1 minutes
  The chest size (in cm) is being recorded.
Patient characteristics - Age | 1 minutes
  The following patient characteristic is being transferred from the clinical internal database (obtained in the CRR on a regular basis): The age of the participant (in years, decimal) is being recorded.
Patient characteristics - Stationary or ambulant | 1 minutes
  The following patient characteristic is being transferred from the clinical internal database (obtained in the CRR on a regular basis): It will be recorded whether the patient is stationary or ambulant.
Patient characteristics - Dominant side | 1 minutes
  The following patient characteristic is being transferred from the clinical internal database (obtained in the CRR on a regular basis): The dominant body side (left or right) is being recorded.
Patient characteristics - Walking aid | 1 minutes
  The following patient characteristic is being transferred from the clinical internal database (obtained in the CRR on a regular basis):
  If applicable: The type of walking aid (open-ended question) is being recorded.
Patient characteristics - Six minute walking test | 1 minutes
  The following patient characteristic is being transferred from the clinical internal database (obtained in the CRR on a regular basis): Upon availability the outcome of the Six-minute walking test will be recorded (distance in meters. Longer distance corresponds to a better outcome.).
Patient characteristics - BAECKE score | 1 minutes
  The following patient characteristic is being transferred from the clinical internal database (obtained in the CRR on a regular basis): BAECKE physical activity questionnaire (Score between 0: no activity, and 10: high activity).
Patient characteristics - Fugl-Meyer score | 1 minutes
  The following patient characteristic is being transferred from the clinical internal database (obtained in the CRR on a regular basis): Lower limb subset of the Fugl-Meyer score. Fugl-Meyer assessment measures the sensorimotor function. (Score between 0: no function and 34: full functionality).

CONTACTS AND LOCATIONS:
Overall Officials: Urs Keller, PhD, Principal Investigator — Ecole Polytechnique Fédérale de Lausanne
Locations (1):
- Clinique Romande de Réadaptation (CRR), SUVAcare, Sion, Valais, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Freund P, Weiskopf N, Ward NS, Hutton C, Gall A, Ciccarelli O, Craggs M, Friston K, Thompson AJ. Disability, atrophy and cortical reorganization following spinal cord injury. Brain. 2011 Jun;134(Pt 6):1610-22. doi: 10.1093/brain/awr093. Epub 2011 May 17. PMID 21586596
- [Background] Kennedy P, Rogers BA. Anxiety and depression after spinal cord injury: a longitudinal analysis. Arch Phys Med Rehabil. 2000 Jul;81(7):932-7. doi: 10.1053/apmr.2000.5580. PMID 10896007
- [Background] Fehr L, Langbein WE, Skaar SB. Adequacy of power wheelchair control interfaces for persons with severe disabilities: a clinical survey. J Rehabil Res Dev. 2000 May-Jun;37(3):353-60. PMID 10917267
- [Background] Hunt PC, Boninger ML, Cooper RA, Zafonte RD, Fitzgerald SG, Schmeler MR. Demographic and socioeconomic factors associated with disparity in wheelchair customizability among people with traumatic spinal cord injury. Arch Phys Med Rehabil. 2004 Nov;85(11):1859-64. doi: 10.1016/j.apmr.2004.07.347. PMID 15520982
- [Background] Meyns P, Van de Crommert HW, Rijken H, van Kuppevelt DH, Duysens J. Locomotor training with body weight support in SCI: EMG improvement is more optimally expressed at a low testing speed. Spinal Cord. 2014 Dec;52(12):887-93. doi: 10.1038/sc.2014.172. Epub 2014 Oct 14. PMID 25311847
- [Background] Crompton S, Khemlani M, Batty J, Ada L, Dean C, Katrak P. Practical issues in retraining walking in severely disabled patients using treadmill and harness support systems. Aust J Physiother. 2001;47(3):211-3. doi: 10.1016/s0004-9514(14)60268-3. No abstract available. PMID 11552877
- [Background] Wessels M, Lucas C, Eriks I, de Groot S. Body weight-supported gait training for restoration of walking in people with an incomplete spinal cord injury: a systematic review. J Rehabil Med. 2010 Jun;42(6):513-9. doi: 10.2340/16501977-0525. PMID 20549154
- [Background] Dobkin B, Barbeau H, Deforge D, Ditunno J, Elashoff R, Apple D, Basso M, Behrman A, Harkema S, Saulino M, Scott M; Spinal Cord Injury Locomotor Trial Group. The evolution of walking-related outcomes over the first 12 weeks of rehabilitation for incomplete traumatic spinal cord injury: the multicenter randomized Spinal Cord Injury Locomotor Trial. Neurorehabil Neural Repair. 2007 Jan-Feb;21(1):25-35. doi: 10.1177/1545968306295556. PMID 17172551
- [Background] Franceschini M, Carda S, Agosti M, Antenucci R, Malgrati D, Cisari C; Gruppo Italiano Studio Allevio Carico Ictus. Walking after stroke: what does treadmill training with body weight support add to overground gait training in patients early after stroke?: a single-blind, randomized, controlled trial. Stroke. 2009 Sep;40(9):3079-85. doi: 10.1161/STROKEAHA.109.555540. Epub 2009 Jun 25. PMID 19556526
- [Background] Hoyer E, Jahnsen R, Stanghelle JK, Strand LI. Body weight supported treadmill training versus traditional training in patients dependent on walking assistance after stroke: a randomized controlled trial. Disabil Rehabil. 2012;34(3):210-9. doi: 10.3109/09638288.2011.593681. PMID 21954995
- [Background] Ada L, Dean CM, Hall JM, Bampton J, Crompton S. A treadmill and overground walking program improves walking in persons residing in the community after stroke: a placebo-controlled, randomized trial. Arch Phys Med Rehabil. 2003 Oct;84(10):1486-91. doi: 10.1016/s0003-9993(03)00349-6. PMID 14586916
- [Background] Kosak MC, Reding MJ. Comparison of partial body weight-supported treadmill gait training versus aggressive bracing assisted walking post stroke. Neurorehabil Neural Repair. 2000;14(1):13-9. doi: 10.1177/154596830001400102. PMID 11228945
- [Background] Visintin M, Barbeau H, Korner-Bitensky N, Mayo NE. A new approach to retrain gait in stroke patients through body weight support and treadmill stimulation. Stroke. 1998 Jun;29(6):1122-8. doi: 10.1161/01.str.29.6.1122. PMID 9626282
- [Background] Teixeira da Cunha Filho I, Lim PA, Qureshy H, Henson H, Monga T, Protas EJ. A comparison of regular rehabilitation and regular rehabilitation with supported treadmill ambulation training for acute stroke patients. J Rehabil Res Dev. 2001 Mar-Apr;38(2):245-55. PMID 11392657
- [Background] Werner C, Von Frankenberg S, Treig T, Konrad M, Hesse S. Treadmill training with partial body weight support and an electromechanical gait trainer for restoration of gait in subacute stroke patients: a randomized crossover study. Stroke. 2002 Dec;33(12):2895-901. doi: 10.1161/01.str.0000035734.61539.f6. PMID 12468788
- [Background] Nilsson L, Carlsson J, Danielsson A, Fugl-Meyer A, Hellstrom K, Kristensen L, Sjolund B, Sunnerhagen KS, Grimby G. Walking training of patients with hemiparesis at an early stage after stroke: a comparison of walking training on a treadmill with body weight support and walking training on the ground. Clin Rehabil. 2001 Oct;15(5):515-27. doi: 10.1191/026921501680425234. PMID 11594641
- [Background] Sullivan KJ, Brown DA, Klassen T, Mulroy S, Ge T, Azen SP, Winstein CJ; Physical Therapy Clinical Research Network (PTClinResNet). Effects of task-specific locomotor and strength training in adults who were ambulatory after stroke: results of the STEPS randomized clinical trial. Phys Ther. 2007 Dec;87(12):1580-602. doi: 10.2522/ptj.20060310. Epub 2007 Sep 25. PMID 17895349
- [Background] Mackay-Lyons M, McDonald A, Matheson J, Eskes G, Klus MA. Dual effects of body-weight supported treadmill training on cardiovascular fitness and walking ability early after stroke: a randomized controlled trial. Neurorehabil Neural Repair. 2013 Sep;27(7):644-53. doi: 10.1177/1545968313484809. Epub 2013 Apr 18. PMID 23599221
- [Background] Combs-Miller SA, Kalpathi Parameswaran A, Colburn D, Ertel T, Harmeyer A, Tucker L, Schmid AA. Body weight-supported treadmill training vs. overground walking training for persons with chronic stroke: a pilot randomized controlled trial. Clin Rehabil. 2014 Sep;28(9):873-84. doi: 10.1177/0269215514520773. Epub 2014 Feb 11. PMID 24519922
- [Background] Combs SA, Dugan EL, Ozimek EN, Curtis AB. Effects of body-weight supported treadmill training on kinetic symmetry in persons with chronic stroke. Clin Biomech (Bristol). 2012 Nov;27(9):887-92. doi: 10.1016/j.clinbiomech.2012.06.011. Epub 2012 Jul 17. PMID 22809736
- [Background] Burgess JK, Weibel GC, Brown DA. Overground walking speed changes when subjected to body weight support conditions for nonimpaired and post stroke individuals. J Neuroeng Rehabil. 2010 Feb 11;7:6. doi: 10.1186/1743-0003-7-6. PMID 20149244
- [Background] Lamontagne A, Fung J. Faster is better: implications for speed-intensive gait training after stroke. Stroke. 2004 Nov;35(11):2543-8. doi: 10.1161/01.STR.0000144685.88760.d7. Epub 2004 Oct 7. PMID 15472095
- [Background] Sousa CO, Barela JA, Prado-Medeiros CL, Salvini TF, Barela AM. The use of body weight support on ground level: an alternative strategy for gait training of individuals with stroke. J Neuroeng Rehabil. 2009 Dec 1;6:43. doi: 10.1186/1743-0003-6-43. PMID 19951435
- [Background] Swinnen E, Baeyens JP, Pintens S, Van Nieuwenhoven J, Ilsbroukx S, Clijsen R, Buyl R, Goossens M, Meeusen R, Kerckhofs E. Trunk muscle activity during walking in persons with multiple sclerosis: the influence of body weight support. NeuroRehabilitation. 2014;34(2):323-35. doi: 10.3233/NRE-131044. PMID 24419023
- [Background] Pennycott A, Vallery H, Wyss D, Spindler M, Dewarrat A, Riener R. A novel body weight support system extension: initial concept and simulation study. IEEE Int Conf Rehabil Robot. 2013 Jun;2013:6650489. doi: 10.1109/ICORR.2013.6650489. PMID 24187306
- [Background] Winter DA, MacKinnon CD, Ruder GK, Wieman C. An integrated EMG/biomechanical model of upper body balance and posture during human gait. Prog Brain Res. 1993;97:359-67. doi: 10.1016/s0079-6123(08)62295-5. PMID 8234761
- [Background] van den Brand R, Heutschi J, Barraud Q, DiGiovanna J, Bartholdi K, Huerlimann M, Friedli L, Vollenweider I, Moraud EM, Duis S, Dominici N, Micera S, Musienko P, Courtine G. Restoring voluntary control of locomotion after paralyzing spinal cord injury. Science. 2012 Jun 1;336(6085):1182-5. doi: 10.1126/science.1217416. PMID 22654062
- [Background] Awai L, Bolliger M, Ferguson AR, Courtine G, Curt A. Influence of Spinal Cord Integrity on Gait Control in Human Spinal Cord Injury. Neurorehabil Neural Repair. 2016 Jul;30(6):562-72. doi: 10.1177/1545968315600524. Epub 2015 Oct 1. PMID 26428035
- [Background] Straube DD, Holleran CL, Kinnaird CR, Leddy AL, Hennessy PW, Hornby TG. Effects of dynamic stepping training on nonlocomotor tasks in individuals poststroke. Phys Ther. 2014 Jul;94(7):921-33. doi: 10.2522/ptj.20130544. Epub 2014 Mar 13. PMID 24627428
- [Background] von Zitzewitz J, Asboth L, Fumeaux N, Hasse A, Baud L, Vallery H, Courtine G. A neurorobotic platform for locomotor prosthetic development in rats and mice. J Neural Eng. 2016 Apr;13(2):026007. doi: 10.1088/1741-2560/13/2/026007. Epub 2016 Feb 10. PMID 26860920
- [Background] Dominici N, Keller U, Vallery H, Friedli L, van den Brand R, Starkey ML, Musienko P, Riener R, Courtine G. Versatile robotic interface to evaluate, enable and train locomotion and balance after neuromotor disorders. Nat Med. 2012 Jul;18(7):1142-7. doi: 10.1038/nm.2845. PMID 22653117
- [Background] Wenger N, Moraud EM, Raspopovic S, Bonizzato M, DiGiovanna J, Musienko P, Morari M, Micera S, Courtine G. Closed-loop neuromodulation of spinal sensorimotor circuits controls refined locomotion after complete spinal cord injury. Sci Transl Med. 2014 Sep 24;6(255):255ra133. doi: 10.1126/scitranslmed.3008325. PMID 25253676
- [Background] Vallery H, Lutz P, von Zitzewitz J, Rauter G, Fritschi M, Everarts C, Ronsse R, Curt A, Bolliger M. Multidirectional transparent support for overground gait training. IEEE Int Conf Rehabil Robot. 2013 Jun;2013:6650512. doi: 10.1109/ICORR.2013.6650512. PMID 24187327
- [Background] Swinnen E, Baeyens JP, Pintens S, Van Nieuwenhoven J, Ilsbroukx S, Buyl R, Ron C, Goossens M, Meeusen R, Kerckhofs E. Trunk kinematics during walking in persons with multiple sclerosis: the influence of body weight support. NeuroRehabilitation. 2014;34(4):731-40. doi: 10.3233/NRE-141089. PMID 24796441
- [Background] Ganesan M, Sathyaprabha TN, Gupta A, Pal PK. Effect of partial weight-supported treadmill gait training on balance in patients with Parkinson disease. PM R. 2014 Jan;6(1):22-33. doi: 10.1016/j.pmrj.2013.08.604. Epub 2013 Sep 8. PMID 24021298
- [Background] Miyai I, Fujimoto Y, Yamamoto H, Ueda Y, Saito T, Nozaki S, Kang J. Long-term effect of body weight-supported treadmill training in Parkinson's disease: a randomized controlled trial. Arch Phys Med Rehabil. 2002 Oct;83(10):1370-3. doi: 10.1053/apmr.2002.34603. PMID 12370870
- [Background] Threlkeld AJ, Cooper LD, Monger BP, Craven AN, Haupt HG. Temporospatial and kinematic gait alterations during treadmill walking with body weight suspension. Gait Posture. 2003 Jun;17(3):235-45. doi: 10.1016/s0966-6362(02)00105-4. PMID 12770637
- [Background] Dragunas AC, Gordon KE. Body weight support impacts lateral stability during treadmill walking. J Biomech. 2016 Sep 6;49(13):2662-2668. doi: 10.1016/j.jbiomech.2016.05.026. Epub 2016 Jun 1. PMID 27282960
- [Background] Lewek MD. The influence of body weight support on ankle mechanics during treadmill walking. J Biomech. 2011 Jan 4;44(1):128-33. doi: 10.1016/j.jbiomech.2010.08.037. Epub 2010 Sep 19. PMID 20855074
- [Background] Mignardot JB, Le Goff CG, van den Brand R, Capogrosso M, Fumeaux N, Vallery H, Anil S, Lanini J, Fodor I, Eberle G, Ijspeert A, Schurch B, Curt A, Carda S, Bloch J, von Zitzewitz J, Courtine G. A multidirectional gravity-assist algorithm that enhances locomotor control in patients with stroke or spinal cord injury. Sci Transl Med. 2017 Jul 19;9(399):eaah3621. doi: 10.1126/scitranslmed.aah3621. PMID 28724575